CLINICAL TRIAL: NCT00295724
Title: A Multi-Center, Double-Blind, Placebo-Controlled Randomized Study of Bicifadine 200 mg BID in the Treatment of Chronic Low Back Pain
Brief Title: Efficacy and Safety of Bicifadine in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DOV Pharmaceutical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOV-075-021
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Low Back Pain
Keywords: bicifadine; chronic low back pain
MeSH Terms: interventions — bicifadine

INTERVENTIONS:
Drug: Bicifadine

SUMMARY:
* The primary objectives of this placebo-controlled clinical trial are to evaluate the analgesic efficacy and safety of bicifadine 200 mg BID compared with placebo in patients with moderate to severe chronic low back pain.
* The secondary objectives are to evaluate the effect of bicifadine on function and general quality of life, to evaluate safety following discontinuation of bicifadine treatment and to investigate the population pharmacokinetics of bicifadine.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with low back pain assessed as Class 1, Class 2 or Class 3 according to the Quebec Task Force Classification for Spinal Disorders and without detectable leg weakness on neurological examination.
* Patients with pain categorized as Class 1 according to the Quebec Task Force Classification must have a Roland-Morris Disability Rating of >17 at baseline to qualify. Patients with pain categorized as Class 2 or Class 3 according to the Quebec Task Force Classification must have a Roland-Morris Disability Rating of at least 10 at baseline to qualify.
* Patients must have required daily analgesics for the treatment of low back pain for at least 3 months prior dosing.

Main Exclusion Criteria:

* Patients may not have persistent moderate or severe pain in a location other than the lower back (with the exception of radiation to the lower extremity).
* Patients must not have had lower back surgery within 6 months prior to baseline, nor epidural corticosteroid injections within 3 months prior to baseline.
* Patients may not have an unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-10

PRIMARY OUTCOMES:
Pain Severity Rating (100 mm visual analog scale)

SECONDARY OUTCOMES:
Short-Form McGill Pain Questionnaire (SF-MPQ)
Roland-Morris Disability Questionnaire (RDQ)
Short-Form 36 (SF-36) Health Survey
Patient's Global Impression of Change (7-point categorical scale)